CLINICAL TRIAL: NCT02714114
Title: Collection of First-void Urine Samples for the Development of Standard Operating Procedures for Anti-HPV (Human Papillomavirus) Antibody Detection in First-void Urine: the AB-SOP Study
Brief Title: Standard Operating Procedures for Anti-HPV (Human Papillomavirus) Antibody Detection in First-void Urine (AB-SOP Study)
Acronym: AB-SOP
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Professor Pierre Van Damme, MD, PhD, Universiteit Antwerpen
Other Study IDs: B300201525584
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Human Papilloma Virus Infection
Keywords: Antibodies; Vaccination; Self-sampling; First-void urine; Serum
MeSH Terms: conditions — Papillomavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples and Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: HPV vaccinated group: Women (18-26 years old) whom are previously vaccinated with the bivalent (Cervarix) or quadrivalent (Gardasil) prophylactic HPV vaccine.
  No clinical evaluations will be performed.
  Interventions: Other: First-void urine collection; Other: Blood draw
- Controls: HPV unvaccinated group: Women (18-26 years old) whom are not vaccinated with the bivalent (Cervarix) or quadrivalent (Gardasil) prophylactic HPV vaccine.
  No clinical evaluations will be performed.
  Interventions: Other: First-void urine collection; Other: Blood draw

INTERVENTIONS:
Other: First-void urine collection — One time collection of ca. 20ml of first-void urine (i.e. the initial stream of the urine void) with the Colli-PeeTM device (Novosanis).
  Other Names: FV urine
Other: Blood draw — One time blood sample collection (5-10 cc) by a study nurse of Centre for the Evaluation of Vaccinations (CEV).
  Other Names: Blood

SUMMARY:
The aim of the study is to develop robust analytical protocols for first-void urine sample preparation and antibody assays to monitor natural and/or vaccine induced immunity against HPV (Human Papillomavirus).

DETAILED DESCRIPTION:
In total 57 women will be included in this trial: 38 vaccinated with an prophylactic HPV vaccine and 19 not vaccinated with a prophylactic HPV vaccine. These women are asked to collect a first-void urine sample with the Colli-PeeTM device (Novosanis). Hereafter, a blood sample of 5-10 cc is collected. The collected urine and blood samples will be used for the development and optimisation of robust analytical protocols for sample preparation and antibody assays.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-26 year
* Cases (n=38): healthy women, fully vaccinated, i.e. receiving all three doses of the bivalent (Cervarix®) or quadrivalent (Gardasil®) HPV vaccine (according to the KCE (Belgian Knowledge Centre for Health) recommendations: age at first vaccination between 10-25 years for the bivalent and 9-26 years for the quadrivalent vaccine).
* Cases should be able to prove their vaccination (brand and schedule) with an official document.
* Control group (n=19): healthy women, self-reported to be not previously vaccinated with a single dose of any prophylactic HPV vaccine available (Gardasil®, Cervarix®, Gardasil-9®)
* Signing informed consent form (ICF).
* Giving consent to the research team (CEV) to contact his/her general practioner and/or gynaecologist to access details of the participants HPV vaccination (schedule) and results of cervical smears/cytology, HPV tests, colposcopy, and biopsy (included in ICF).

Exclusion Criteria:

* Participating in another clinical study at the same time of participating in this study.
* Not able to understand the information brochure/what the study is about
* Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In total 57 women will be included in this trial. During their study visit, participants are asked to collect a first-void urine sample with the Colli-PeeTM device. Hereafter, a blood sample of 5-10 cc is collected. Following sample collection, women are asked to fill in a questionnaire.
  For this pilot study, our study population is based on unequal groups with twice as many cases (vaccinated women) then controls (non-vaccinated women) (k = 2) because our focus is to develop analytical protocols and assays for anti HPV antibodies. This results in a total sample size of 57, including 19 controls (non-vaccinated women) and 38 cases (vaccinated women).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Concentration HPV specific IgG (Immunoglobulin G) in paired first-void urine and serum samples | Within 6 months after study completion
  To detect HPV specific IgG concentrations (ratio HPV specific IgG/total human IgG), in paired first-void urine and serum samples from 57 women to monitor the immune response after vaccination with a prophylactic HPV vaccine (Gardasil or Cervarix).

SECONDARY OUTCOMES:
Concentration HPV specific IgA (Immunoglobulin A) in paired first-void urine and serum samples | Within 6 months after study completion
  To detect HPV specific IgA concentrations (ratio HPV specific IgA/total human IgA), in paired first-void urine and serum samples from 57 women to monitor the immune response after vaccination with a prophylactic HPV vaccine (Gardasil or Cervarix).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Pierre Van Damme, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Keer S, Willhauck-Fleckenstein M, Pattyn J, Butt J, Tjalma WAA, Van Ostade X, Hens N, Van Damme P, Waterboer T, Vorsters A. First-void urine as a non-invasive liquid biopsy source to detect vaccine-induced human papillomavirus antibodies originating from cervicovaginal secretions. J Clin Virol. 2019 Aug;117:11-18. doi: 10.1016/j.jcv.2019.05.004. Epub 2019 May 11. PMID 31129514